CLINICAL TRIAL: NCT04086888
Title: Real World Study of Immune Checkpoint Inhibitors for Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Sun Yat-sen University
Other Study IDs: RWS-ICI-GC
Record Dates: First submitted 2019-09-06; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
Keywords: Immune checkpoint inhibitors
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gastric cancer ranks as the fifth most common and the third most common cause of cancer deaths in the world. In spite of the progresses made in the diagnosis and treatment of gastric cancer in the past decades, the prognosis is still unsatisfied mainly due to recurrence and distant metastasis. Surgical treatment is the first choice for the treatment of early gastric cancer, but it is prone to recurrence and metastasis after surgery. There are relatively few chemotherapy drugs for gastric cancer. Studies have shown that about 13% of gastric cancers have HER2 gene amplification, and there are no other known driver gene other than HER-2. At present, the targeted therapeutic drugs approved for gastric cancer in China are only trastuzumab and apatinib.

Immune checkpoint inhibitors, including PD-1 inhibitors, PD-L1 inhibitors and CTLA-4 inhibitors, have achieved significant therapeutic effects in a variety of tumors and are expected to alter the current state of treatment of tumors. In gastric cancer, the KEYNOTE-012 study demonstated the efficacy of Pembrolizumab in patients with PD-L1 positive advanced gastric cancer. The study showed that 53% of patients had tumor retraction, and 22% achieved partial imaging remission with a median duration of 40 weeks. At the same time, Pembrolizumab is also less toxic than standard second-line chemotherapy. However, Are the Immune checkpoint inhibitors should be used as single-drug or in combination with chemotherapy? Are the Immune checkpoint inhibitors should be used in the first-line or in the back-line? And which is the best combination therapy? For these issues, there is no conclusion yet.

This observational study included all patients with gastric cancer who used Immune checkpoint inhibitors in clinical practice, regardless of treatment lines and combination with different chemotherapy. Through follow-up observations, the aim of this study is to analyze the efficacy of Immune checkpoint inhibitors for gastric cancer in the real world, and to explore the differences in the efficacy of Immune checkpoint inhibitors in different stages of treatment, as well as the efficacy of different chemotherapy combinations, so as to provide clinical evidence for the use of immunotherapy for advanced gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age above 16, male or female.
2. patients with gastric cancer confirmed by pathology through tumor biopsy or puncture tissue.
3. the patient was assessed as untreatable by surgery.
4. patients received first line, second-line or third-line chemotherapy and were treated with immunne checkpoint inhibitors.
5. the patient had complete preliminary pathological information, tumor site, pathological type and other information.
6. the patient must have adequate tumor tissue or 5-10 FFPE white tablets to provide; After treatment, patients were returned to the hospital for re-examination every 3 treatment cycles, and plasma and peripheral blood samples could be obtained during the whole process.
7. other indicators of the patients met the general clinical trial enrollment conditions.
8. subjects read and fully understand the instructions to patients, and sign the informed consent.

   -

Exclusion Criteria:

1. Patients who cannot provide peripheral blood samples prior treatment.
2. Patients with severe infection will be excluded.
3. Patients with other serious disease besides gastric cancer will be excluded.
4. Pregnant women will be excluded.
5. Patients who are alcoholic or drug abusers will be excluded.
6. Patients with a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data will be excluded.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 170 patients with advanced gastric cancer were enrolled. Patients need to be treated with immunocheckpoint inhibitors or immunocheckpoint inhibitors in combination with chemotherapy. 10ml of edta-anticoagulant blood was collected before the first treatment of the enrolled patients, and the blood samples were gently reversed in the anticoagulant tube for several times to fully anticoagulate. The upper plasma and the lower blood cells were centrifuged at 1800g for 10 min within 4 hours, respectively, and stored at -80 ℃ for later use and provide 10-15 tumor tissue white sheets.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2019-12-17 (Estimated); Study Completion 2020-06-20 (Estimated)

PRIMARY OUTCOMES:
OS (overall survival) | through study completion, an average of 3 years
  the time from receiving the first dose of Immune checkpoint Inhibitors treatment to death or the end of the observation

SECONDARY OUTCOMES:
progression-free survival (PFS) | through study completion, an average of 3 years
  the time from receiving the first dose of Immune checkpoint Inhibitors treatment to progression of disease (PD) or death

CONTACTS AND LOCATIONS:
Overall Officials: Rui-hua Xu, MD, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided